CLINICAL TRIAL: NCT03000062
Title: Treatment of Overweight in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik L Werner, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDN01
Record Dates: First submitted 2016-12-13; First posted 2016-12-21 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Overweight and Obesity; Nutritional and Metabolic Diseases
Keywords: overweight, general practice
MeSH Terms: conditions — Overweight; Obesity; Nutritional and Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Participant
Masking Description: ID of participating patients are only available through the participating Family phyisican
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): 12 Family physicians in primary care will constitute the Intervention group. They will enroll 10 patients each from their ordinary practice. The physicians will be provided with a specific course on the treatment model of the study, including how to collect and register data. They will have a detailed manual indicating the content of each visit.
  Following recruitment and consent, the patient will meet for the first visit in the study one week later. At this visit the patient will be provided with detailed information on the content and preparation for all meals. Data will be collected.
  The manual describes a diet in accordance with official guidelines providing the patient 1600Kcal per day.
  The following visits will take place after 4 weeks, 8 weeks, 4 months, 8 months and 12 months from the first visit. Data will be collected at all visits, and also at 6 and 12 months follow-up.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): 12 Family physicians in primary care will constitute the Control group. They will enroll 10 patients each from their ordinary practice. The physicians will not be provided with any information of the treatment model of the study but they will have all information about how to collect and register data.
  The patients on this group will also sign consent to provide data and therefore they will know about the study but they do not get any specific information about weight loss other than the general information that their physician may tell them.
  The patients in the Control Group will be asked to give data on inclusion visit and again 12 months later, and also at 6 and 12 months thereafter (i.e. 0, 12, 18 and 24 months from inclusion).

INTERVENTIONS:
Behavioral: Intervention group — Please see the preceding section
  Arms: Intervention group

SUMMARY:
In this study the investigators want to explore the feasibility and effect of a simple intervention provided by primary care physicians on treatment for overweight in general practice. Regular patients visiting their ordinary family physician will be asked for participation if they comply with the inclusion criteria. If so, they will follow a detailed food list for 12 months with regular visits to the doctor. At each visit, the participating patients will be asked about their progress on weight loss and all measurements will be made. Simultaneously a control group of primary care physicians will also recruit patients that fulfill the inclusion criteria. These patients will also provide data that will serve as Control to the intervention group.

DETAILED DESCRIPTION:
The number of patients with overweight is increasing and a daily issue in general practice. Many patients wish to discuss their weight problem with their family physician but many of these feel helpless to guide their patients in how to reduce weight. Providing useful and correct information should not be so difficult but many doctors choose to refer their patients to dietary courses or follow-up in specialist health care.In this study the investigators wish to implement a simple tool for treatment of overweight in primary care by providing the patients a detailed list for all meals that will ensure a weight loss. The patients will be given a close follow-up by their doctor, and the motivating conversation and list of meals will be the only treatment given.

The study is a cluster randomised controlled trial where all general practices in the area of Moss city in Norway will be asked to participate. Half of the physicians will constitute the intervention group while the other half will serve as control group. Each participating doctor in both groups will recruit patients according to the eligibility criteria. The doctors in the intervention group will be provided with a course to learn the intervention and have a manual to follow for each patient. All participating patients of both groups will be asked to meet regularly for data collection.

According to the power calculation, a number of 12 physicians in each group will be sufficient if they recruit 10 patients each.

The intervention will be conducted for 12 months and thereafter data will be continued to be collected at 6 and 12 months after.

ELIGIBILITY:
Inclusion Criteria:

* BMI _> 30 OR _25 With at least one Medical condition related to overweight (hypertension, dyslipidemia, metabolic syndrome, diabetes mellitus II, hip- or knee pain)
* written consent
* sufficient knowledge in Norwegian Language to acquire the written and oral information

Exclusion Criteria:

* any ongoing cancer condition
* any current medication impacting on weight

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Weight reduction | 12 months
  10% weight reduction measured as kilo weight at inclusion

SECONDARY OUTCOMES:
Blood pressure | 12 months
  Blood pressure measured as mean of three measurements at rest
HbA1c | 12 months
  Blood samples
Waist measure | 12 months
  Any reduction in cm of waist measure
Total Cholesterol | 12 months
  Blood samples

OTHER OUTCOMES:
Qualitative study | 24 months
  Participating physicians and patients will be interviewed about their experiences With the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jørund Straand, Prof., Ph.D, Study Director — University of Oslo

IPD SHARING:
Plan to Share IPD: Undecided
Data on all outcomes will be available to researchers on request

REFERENCES:
- [Derived] Nilsen MD, Mdala I, Werner EL. Treatment of overweight and obesity in general practice: a cluster randomised trial. BMJ Nutr Prev Health. 2023 Nov 29;6(2):326-331. doi: 10.1136/bmjnph-2023-000721. eCollection 2023. PMID 38618545